CLINICAL TRIAL: NCT04437862
Title: A Prospective, Multi-Center, Single Arm Study to Evaluate the Q Revascularization System for Neurointervention in Acute Ischemic Stroke: The EvaQ Study
Brief Title: A Study to Evaluate the Q Revascularization System for Neurointervention in Acute Ischemic Stroke
Acronym: EvaQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MIVI Neuroscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 101773
Record Dates: First submitted 2020-06-16; First posted 2020-06-18 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Acute Stroke; Cerebral Ischemia
MeSH Terms: conditions — Stroke; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Q Revascularization System (Experimental)
  Interventions: Device: Q Revascularization System

INTERVENTIONS:
Device: Q Revascularization System — Q Revascularization System for mechanical thrombectomy

SUMMARY:
Assess the safety and efficacy of the Q Revascularization System to remove thrombi and emboli from the neurovasculature in patients experiencing an acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Pre-stroke independent functional status in activities of daily living with mRS 0-1.
* A disabling stroke defined as NIHSS ≥ 6
* In USA thrombolytic therapy (IV tPA) received within 3 hours of onset/ last known well, in Europe treatment with IV tPA received within 4.5 hours from onset/ last known well OR ineligibility for thrombolytic therapy
* Endovascular treatment intended to be initiated < 8 hours from onset of symptoms or last known well time
* Confirmed symptomatic large vessel occlusion of the intracranial internal carotid artery, middle cerebral artery, M1, M2, basilar or intracerebral vertebral artery by baseline neuroimaging CTA/MRA and angiographic imaging with a mTICI Score 0-1
* For strokes in the anterior circulation the following imaging criteria should also be met: MRI criterion of volume of diffusion restriction visually assessed ≤50 mL OR CT criterion of ASPECTS 6 to 10 on baseline CT or CTA-source images or, significantly lowered cerebral blood volume (CBV) ≤50 mL
* For strokes in the basilar or vertebral artery, the following imaging criterion should also be met: pc-ASPECTS score 8 to 10 on baseline CT, CTA-source images, or MRI
* Signed informed consent from subject, acceptable person responsible (e.g. LAR) and/or according to County specific regulatory requirements and local ethical committee or review board requirements

Exclusion Criteria:

* CT or MRI evidence of intracranial hemorrhage on presentation
* CT or MRI showing mass effect or intracranial tumor (meningioma > 2 cm in diameter).
* Previous stroke within the past 3 months
* Rapidly improving neurological status as determined by Investigator/Neurologist
* Renal failure/insufficiency with >3.0 mg/dL creatinine prior to procedure
* Severe, sustained hypertension resistant to treatment (SBP >185 mmHg or DBP >110 mmHg)
* Use of warfarin anticoagulation with International Normalized Ratio (INR) > 3.0 at the time of the procedure or any known hemorrhagic or coagulation deficiency
* For patients who have received a direct thrombin inhibitor within the last 48 hours; partial thromboplastin time (PTT) > 2.0 times the normal prior to procedure
* Platelet count < 50,000 mm3
* Cerebral vasculitis or evidence of active systemic infection
* Suspicion of aortic dissection, presumed septic embolus, or suspicion of bacterial endocarditis
* Clinical symptoms suggestive of bilateral stroke or occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation)
* Seizure due to stroke
* Pregnancy
* Severe contrast allergy or absolute contraindication to iodinated contrast
* Presence of a carotid artery stenosis or occlusion requiring balloon angioplasty or stenting at time of the procedure
* Difficult endovascular access or difficult aortic arch or severe neurovascular tortuosity that will result in an inability to deliver endovascular therapy
* Evidence of dissection in the carotid or target artery for treatment
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic
* Active participation in another study involving an investigational drug or device
* A severe or fatal comorbid illness that will prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient
* Unwillingness to complete follow up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Successful revascularization rate | Procedure end
  Successful revascularization defined at modified Treatment in Cerebral Ischemia (mTICI) 2b-3 at the end of the procedure
Symptomatic intracranial haemorrhage rate | 36 hours post procedure
  Symptomatic intracranial haemorrhage (ICH) as detected by CT/MRI and a clinical deterioration of NIHSS change ≥ 4

SECONDARY OUTCOMES:
Successful revascularization rate with study device | Procedure
  Successful revascularization defined as mTICI 2b-3 flow after all aspiration attempts with the study device
Successful revascularization rate on the first attempt with study device | Procedure
  Successful revascularization defined as mTICI 2b-3 flow after the first aspiration attempt with the study device
Procedure Time | Procedure
  Time from groin puncture to successful revascularization defined as final mTICI 2b-3 flow
ENT rate | Procedure
  Embolization to a new vascular territory (ENT) during procedure
Procedure Complications | Procedure through 90 days
  Rate of procedure related complications
ICH | 36 hours post procedure
  Occurrence of all intracranial hemorrhage using the Heidelberg Bleeding Classification.
Good functional outcome | 90 days post procedure
  Good functional outcome measured by Modified Rankin Score (mRS) defined as a value of 0-2
Mortality | 90 days post procedure
  All cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cognard, PhD, MD, Principal Investigator — Hôpital Purpan; Lucas Elijovich, MD, Principal Investigator — University of Tennessee Health Sciences Center; Brian Jankowitz, MD, Principal Investigator — JFK University Medical Center
Locations (8):
- United States (4):
  - University of South Florida, Tampa, Florida
  - Cooper University Health Care, Camden, New Jersey
  - University at Buffalo Neurosurgery, Buffalo, New York
  - Baptist Memorial Hospital, Memphis, Tennessee
- France (4):
  - CHU Pellegrin, Bordeaux
  - CHU Urbains, Nancy
  - CHU Bicetre Paris, Paris
  - Hôpital Purpan, Toulouse

IPD SHARING:
Plan to Share IPD: No